CLINICAL TRIAL: NCT05496660
Title: The Effect of the Nordic Hamstring Exercise and Kinesio Taping on the Hamstring Strength and Sprint Performance in Collegiate Sprinters
Brief Title: The Effect of NHE and KT on the Hamstring Strength and Sprint Performance in Collegiate Sprinters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin University of Sport (Other)
Responsible Party: Principal Investigator, Wei Zheng, Professor, Tianjin University of Sport
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NHE_KT
Record Dates: First submitted 2022-08-03; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Hamstring Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NHE+KT (Experimental): the Nodic hamstring exercise plus the kinesio taping with tension during 4-week consisting 12 sessions
  Interventions: Other: NHE+KT
- NHE (Sham Comparator): the Nordic hamstring exercise plus taping wihout tension during 4-week consisting 12 sessions
  Interventions: Other: NHE

INTERVENTIONS:
Other: NHE+KT — the Nodic hamstring exercise plus the kinesio taping with tension during 4-week consisting 12 sessions
  Arms: NHE+KT
Other: NHE — the Nodic hamstring exercise plus the kinesio taping without tension during 4-week consisting 12 sessions
  Arms: NHE

SUMMARY:
The invesitgators performed a randomized controlled trial on collegiate sprinters to explore the combined effect of the NHE and KT and randomly allocated the subjects into the experimental (NHE+KT) or control (NHE) group by an independent researcher using the sealed envelopes method.

To calculate the sample size, a Cohen's d effect size of 0.4, an alpha level of 0.05, a test power of 0.95 were configured to G*Power software, at least 34 samples were computed. Considering the dropouts, 40 male collegiate sprinters were enrolled, explained the procedures of this study and voluntarily written informed consent. Inclusion criteria was that participants must be male, aged 18 years or older, training at the university level at least 4 times per week, with no history of lower limb injury within the last 6 months and no previous experience of the NHE or KT. Participants who had lower limb mobility limitation or injury especially HSI within 6 months and associated musculoskeletal, respiratory or cardiovascular diseases and was allergic to kinesio tape were excluded.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be male, aged 18 years or older, training at the university level at least 4 times per week, with no history of lower limb injury within the last 6 months and no previous experience of the NHE or KT.

Exclusion Criteria:

* Participants who had lower limb mobility limitation or injury especially HSI within 6 months and associated musculoskeletal, respiratory or cardiovascular diseases and was allergic to kinesio tape were excluded.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
isokinetic hamstring eccentric peak torque | 4-week
  eccentric peak torque measured by Cybex
30m sprint performance | 4-week
  30m sprint time

SECONDARY OUTCOMES:
Hecc/Qcon Ratio | 4-week
  hamstring eccentric peak torque/Quadriceps concentric peak torque

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin University of Sport, Tianjin, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol